CLINICAL TRIAL: NCT04694768
Title: The Effect of Implementing a Nursing Program Intervention on Improvement of Health Quality of Post Covid-19 Patients
Brief Title: Implementation of Rehabilitation Program for Post COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU19
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Post COVID-19 Syndrome; Rehabilitation
Keywords: nursing program; health quality of life
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Rehabilitation — Rehabilitation program

SUMMARY:
Many people who have suffered from the effects of this disease might now be at risk of long-term impairment and disability. The extent of this impairment and disability is yet unknown, but it is clear from early research that these patients will be in need of rehabilitation in all phases of the disease - acute, post-acute and long-term.

Rehabilitation is defined as "a set of interventions designed to reduce disability and optimize functioning in individuals with health conditions in interaction with their environment." Rehabilitation might very well be a key strategy to reduce the impact of COVID-19 on the health and function of people.

A team work is needed to implement this programs which are essential in all phases to facilitate early discharge, but even more to support and empower patients.

ELIGIBILITY:
Inclusion Criteria:

* Post acute COVID-19 patients

Exclusion Criteria:

* Acute COVID-10
* Non- COVID-19 patients
* Recent myocardial infarction
* Recent pulmonary embolism
* Neurologic diseases

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients recovered from SARs-CoV-2 after 4 weeks
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Optimizing health and functioning outcomes | 6 months
  decrease intensive care acquired weakness
improve recovery and reduce disability | 6 months
  decrease dyspnea, fatigue, anxiety and sleep disturbance

CONTACTS AND LOCATIONS:
Locations (1):
- Aliae AR Mohamed-Hussein, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided